CLINICAL TRIAL: NCT01574573
Title: Impact of Weight Loss on Gastroesophageal Reflux Disease in Overweight and Obese Subjects: a Prospective Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed due to lack of recruitment
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Principal Investigator, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS0054
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: GERD; Obesity
Keywords: Obesity; GERD; Weight loss
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese individuals with weight loss (Experimental): Self support, group sessions
  Interventions: Behavioral: Self support, group sessions
- Obese individuals without weight loss (Experimental): self support, group sessions
  Interventions: Behavioral: Self support, group sessions

INTERVENTIONS:
Behavioral: Self support, group sessions — Self support,group sessions

SUMMARY:
By affecting the gastroesophageal pressure gradient, obesity predisposes to reflux of gastric contents. The investigators hypothesized that the loss of weight will decrease this gradient and as a result decrease the severity and frequency of GERD symptoms. GERD negatively affects health related quality of life. Since loss of weight may decrease gastroesophageal reflux, the investigators hypothesized that it obesity contributes to poor quality of life in GERD subjects and losing weight should also favorably impact and improve quality of life in GERD patients.

DETAILED DESCRIPTION:
The current proposal is a prospective, observational cohort study This study aims to determine the impact of structured weight loss (MOVE program) on GERD symptoms in overweight and obese veterans enrolled in a MOVE program. Successful weight loss will be defined as loss of 10% or higher baseline weight at 6 months follow up. Cases will be defined as subjects who achieved successful weight loss and controls as those who did not. GERD symptoms in subjects who lose weight (cases) will be compared to those with no weight loss (controls). Validated GERQ, RDQ and QOLRAD questionnaires will be used to assess prevalence of GERD symptoms, QOL and impact of weight loss on these symptoms. All MOVE participants will complete a validated GERQ, RDQ and QOLRAD questionnaires at baseline MOVE clinic visit and RDQ and QOLRAD during their follow up visits. Patient's total RDQ scores at baseline and follow up visits will be used to determine change in frequency and severity of GERD symptoms with weight loss, similarly change in the total QOLRAD questionnaire scores from baseline will be used to assess change in HRQOL with weight loss. Apart from information provided in MOVE!23, GERQ, RDQ and QOLRAD questionnaires, relevant information pertaining to obesity and GERD association will be obtained from patient's computerized medical records.

The impact of weight loss on GERD symptoms will be assessed. The impact of weight loss on QOL and GERD medication usage among MOVE participants will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Kansas City Veterans Hospital patient who is enrolled in the MOVE weight loss program
* Patients with a BMI > 25 with associated co-morbid medical conditions such as diabetes, high blood pressure, high cholesterol, arthritis, heart disease, low back pain, sleep apnea, or other obesity associated condition.
* Enrollment in MOVE program is optional for patients with a BMI > 25 with no co-morbid medical conditions.
* Enrollment for patients 70 years or older with BMI > 25 is optional and requires mandatory medical clearance prior to beginning new physical activity and closer nutritional supervision to minimize protein, vitamin and mineral deficiencies.

Exclusion Criteria:

* Active cancer other than non-melanoma skin cancer
* End stage COPD, congestive heart failure
* End stage neurologic disorder (Parkinson's, ALS, MS)
* Long-term care facility resident
* End stage renal disease
* Moderate to severe cognitive impairment (dementia, post-stroke)
* Active psychosis or substance abuse
* AIDS (except asymptomatic HIV infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Impact of Weight loss on GERD symptoms | 48 months

SECONDARY OUTCOMES:
Impact of weight loss on quality of life and GERD symptoms | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City VA Medical Center
Locations (2):
- United States (2):
  - Topeka VA Medical Center, Topeka, Kansas
  - Kansas City VA Medical Center, Kansas City, Missouri

REFERENCES:
- [Background] Dent J, El-Serag HB, Wallander MA, Johansson S. Epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2005 May;54(5):710-7. doi: 10.1136/gut.2004.051821. PMID 15831922
- [Background] Kulig M, Nocon M, Vieth M, Leodolter A, Jaspersen D, Labenz J, Meyer-Sabellek W, Stolte M, Lind T, Malfertheiner P, Willich SN. Risk factors of gastroesophageal reflux disease: methodology and first epidemiological results of the ProGERD study. J Clin Epidemiol. 2004 Jun;57(6):580-9. doi: 10.1016/j.jclinepi.2003.10.010. PMID 15246126
- [Background] McDougall NI, Johnston BT, Kee F, Collins JS, McFarland RJ, Love AH. Natural history of reflux oesophagitis: a 10 year follow up of its effect on patient symptomatology and quality of life. Gut. 1996 Apr;38(4):481-6. doi: 10.1136/gut.38.4.481. PMID 8707073
- [Background] Talley NJ, Fullerton S, Junghard O, Wiklund I. Quality of life in patients with endoscopy-negative heartburn: reliability and sensitivity of disease-specific instruments. Am J Gastroenterol. 2001 Jul;96(7):1998-2004. doi: 10.1111/j.1572-0241.2001.03932.x. PMID 11467624
- [Background] Kulig M, Leodolter A, Vieth M, Schulte E, Jaspersen D, Labenz J, Lind T, Meyer-Sabellek W, Malfertheiner P, Stolte M, Willich SN. Quality of life in relation to symptoms in patients with gastro-oesophageal reflux disease-- an analysis based on the ProGERD initiative. Aliment Pharmacol Ther. 2003 Oct 15;18(8):767-76. doi: 10.1046/j.1365-2036.2003.01770.x. PMID 14535869
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] Nebel OT, Fornes MF, Castell DO. Symptomatic gastroesophageal reflux: incidence and precipitating factors. Am J Dig Dis. 1976 Nov;21(11):953-6. doi: 10.1007/BF01071906. PMID 984016
- [Background] El-Serag HB, Kvapil P, Hacken-Bitar J, Kramer JR. Abdominal obesity and the risk of Barrett's esophagus. Am J Gastroenterol. 2005 Oct;100(10):2151-6. doi: 10.1111/j.1572-0241.2005.00251.x. PMID 16181362
- [Background] El-Serag HB. Time trends of gastroesophageal reflux disease: a systematic review. Clin Gastroenterol Hepatol. 2007 Jan;5(1):17-26. doi: 10.1016/j.cgh.2006.09.016. Epub 2006 Dec 4. PMID 17142109
- [Background] Fisher BL, Pennathur A, Mutnick JL, Little AG. Obesity correlates with gastroesophageal reflux. Dig Dis Sci. 1999 Nov;44(11):2290-4. doi: 10.1023/a:1026617106755. PMID 10573376
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Murray L, Johnston B, Lane A, Harvey I, Donovan J, Nair P, Harvey R. Relationship between body mass and gastro-oesophageal reflux symptoms: The Bristol Helicobacter Project. Int J Epidemiol. 2003 Aug;32(4):645-50. doi: 10.1093/ije/dyg108. PMID 12913045